CLINICAL TRIAL: NCT02582255
Title: A Phase 4 Study to Evaluate the Safety and Immunogenicity of Monovalent Oral Polio Vaccine Type 2 in Healthy IPV-vaccinated Children Aged 1 to 5 Years in Lithuania
Brief Title: A Study to Evaluate the Safety and Immunogenicity of Monovalent OPV2 in Children Aged 1 to 5 Years in Lithuania
Acronym: M3-ABMG
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fidec Corporation (Other)
Collaborators: Bill and Melinda Gates Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: M3-ABMG
Record Dates: First submitted 2015-08-04; First posted 2015-10-21 (Estimated); Results first posted 2019-12-16 (Actual); Last update posted 2020-01-14 (Actual); Status verified 2020-01

CONDITIONS: Poliomyelitis
MeSH Terms: conditions — Poliomyelitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sabin mOPV2 1 dose (Experimental): IPV-vaccinated children to receive 1 dose of SABIN mOPV2 (Group 1)
  Interventions: Biological: Sabin mOPV2
- SABIN mOPV2 2 doses (Experimental): IPV-vaccinated children to receive 2 doses of SABIN mOPV2 (Group 2)
  Interventions: Biological: Sabin mOPV2

INTERVENTIONS:
Biological: Sabin mOPV2 — Polio Sabin™ Mono Two (oral) is a licensed, monovalent, live attenuated poliomyelitis virus vaccine of the Sabin strain Type 2 (P 712, Ch, 2ab), propagated in MRC5 human diploid cells. Each two-drop dose (0.1 mL) contains not less than 105.0 CCID50 of Type 2. Magnesium chloride is used as a stabilizer. Polio Sabin™ Mono Two (Oral) contains trace amounts of neomycin sulphate and polymyxin B sulphate.
  One dose of vaccine (0.1 mL) is contained in two drops which are delivered from the polyethylene dropper supplied with vaccine.
  Other Names: mOPV2

SUMMARY:
A Phase 4 study to evaluate the safety and immunogenicity of monovalent oral polio vaccine type 2 in healthy IPV-vaccinated children aged 1 to 5 years in Lithuania.

DETAILED DESCRIPTION:
Sabin 2 will be withdrawn from routine use globally from April 2016 as per the SAGE recommendations at the time of writing this protocol. After this cessation of OPV2, stockpiles of mOPV2 will be maintained for potential use if necessary in response to a future outbreak. However, there is a risk of cVDPV2 from Sabin 2 in settings of low population immunity. Research is ongoing to develop vaccines that are genetically more stable than the currently available Sabin 2-containing OPVs. To generate data on immunogenicity, safety, and genetic stability on the Sabin 2 vaccine (mOPV2) and as a future comparator for new polio vaccine research after the global switch from tOPV to bOPV, this study with mOPV2 is performed to evaluate safety, immunogenicity (humoral and intestinal) and genetic stability endpoints of mOPV2 in children aged 1 to 5 years for better understanding of the stockpile use of this vaccine, and any potential new polio vaccine with a type 2 component in the future.

ELIGIBILITY:
Inclusion Criteria:

1. 1 to 5 years of age, previously vaccinated with three or four doses of IPV.
2. Healthy without obvious medical conditions that preclude entry of the subject into the study as established by the medical history and physical examination.
3. Written informed consent obtained from 1 or 2 parent(s) or legal guardian(s) as per country regulations.

Exclusion Criteria:

1. Previous vaccination against poliovirus outside the national immunization schedule.
2. Any confirmed or suspected immunosuppressive or known immunodeficient condition including human immunodeficiency virus (HIV) infection.
3. Family history of congenital or hereditary immunodeficiency.
4. Major congenital defects or serious uncontrolled chronic illness (neurologic, pulmonary, gastrointestinal, hepatic, renal, or endocrine).
5. Known allergy to any component of the study vaccines or to any antibiotics.
6. Administration of immunoglobulins and/or any blood products since birth or planned administration during the study period.
7. Acute severe febrile illness at day of vaccination deemed by the Investigator to be a contraindication for vaccination (the child can be included at a later time if within age window and all in/exclusion criteria are met.).
8. Member of the subject's household (living in the same house or apartment unit) has received OPV in the last 3 months.
9. Subject who, in the opinion of the Investigator, is unlikely to comply with the protocol or is inappropriate to be included in the study for the safety or the benefit-risk ratio of the subject.

Ages: 1 Year to 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 100 (Actual)
Dates: Start 2015-11; Primary Completion 2016-07 (Actual); Study Completion 2016-12-22 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Vytautas Usonis, Prof, Principal Investigator — Vilnius University

REFERENCES:
- [Derived] Bandyopadhyay AS, Gast C, Brickley EB, Ruttimann R, Clemens R, Oberste MS, Weldon WC, Ackerman ME, Connor RI, Wieland-Alter WF, Wright P, Usonis V. A Randomized Phase 4 Study of Immunogenicity and Safety After Monovalent Oral Type 2 Sabin Poliovirus Vaccine Challenge in Children Vaccinated with Inactivated Poliovirus Vaccine in Lithuania. J Infect Dis. 2021 Jan 4;223(1):119-127. doi: 10.1093/infdis/jiaa390. PMID 32621741

RESULTS

PARTICIPANT FLOW:
Groups:
- Group 1: IPV-vaccinated children receiving 1 dose of SABIN mOPV2.
- Group 2: IPV-vaccinated children receiving 2 doses of SABIN mOPV2.
Period: Overall Study
Arm/Group | Group 1 | Group 2
Started | 50 | 50
Completed | 50 | 47
Not Completed | 0 | 3
Not completed — Protocol Violation | 0 | 3

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Group 1 | Group 2 | Total
Number analyzed (Participants) | 50 | 50 | 100
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 50 | 50 | 100
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 26 | 19 | 45
  Male | 24 | 31 | 55
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 50 | 50 | 100
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  Lithuania | 50 | 50 | 100

OUTCOME MEASURES:

1. Primary Outcome: SAEs and Severe AEs
Description: Incidence of SAEs and severe AEs grade 3 considered consistent with a causal association to study vaccine throughout the study period in children 1 to 5 years.
Time Frame: 3 months
Population: All participants who received at least one dose of vaccine.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 50 | 47
Participants | 0 | 0
Statistical Analysis 1: Comparison: Group 1 vs Group 2; Test type: Other; p = 0.05, Clopper-Pearson

2. Primary Outcome: Seroprotection Rate of Type 2 Polio Neutralizing Antibodies.
Description: Seroprotection rate at type 2 polio neutralizing antibodies measured at D28 after the first dose of mOPV2.
Time Frame: 1 month
Population: All participants who received two doses of vaccines.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 50 | 47
Participants | 50 | 47
Statistical Analysis 1: Comparison: Group 1 vs Group 2; Test type: Other; p = 0.025, Clopper-Pearson

3. Secondary Outcome: Seroprotection Rate for Type 2 Polio Neutralizing Antibodies.
Description: Seroprotection rate for type 2 polio neutralizing antibodies measured at D 28 after the secon dose of mOPV2.
Time Frame: 3 months
Population: All subjects receiving two doses of vaccine.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 2
Number analyzed (Participants) | 47
Participants | 47
Statistical Analysis 1: Comparison: Group 2; Test type: Other; p = 0.025, Clopper-Pearson

4. Secondary Outcome: Incidence of Any Serious Adverse Events (SAEs), Any Solicited AEs, Any Unsolicited AEs, and Any Important Medical Events (IMEs).
Description: Incidence, severity and relationship) of any serious adverse events (SAEs), any solicited AEs, any unsolicited AEs, and any Important Medical Events (IMEs) with the exception of severe related AEs. (primary objective), as well as any laboratory deviations of one or two doses of SABIN mOPV2 in healthy IPV-vaccinated children aged 1 to 5 years.
Time Frame: 3 months
Population: All subjects receiving at least one dose of vaccine.
Measure: Count of Participants; unit: Participants
Arm/Group | Group 1 | Group 2
Number analyzed (Participants) | 50 | 47
Participants | 6 | 9
Statistical Analysis 1: Comparison: Group 1 vs Group 2; Test type: Other; p = 0.05, Clopper-Pearson

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Group 1 | Group 2
All-Cause Mortality (participants affected / at risk) | 0/50 | 0/50
Serious Adverse Events (participants affected / at risk) | 0/50 | 1/50
Other Adverse Events (participants affected / at risk) | 6/50 | 12/50
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 (N=50) | Group 2 (N=50)
Bronchitis (Respiratory, thoracic and mediastinal disorders) | NA | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Group 1 (N=50) | Group 2 (N=50)
Appetite lost (General disorders) | 1 (1) | 0 (0)
Abnormal crying (General disorders) | 1 (1) | 0 (0)
Fever (General disorders) | 0 (0) | 1 (1)
Irritability (General disorders) | 1 (1) | 1 (1)
Vomiting (Gastrointestinal disorders) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 1 (2) | 2 (3)
Bronchitis (Infections and infestations) | 1 (1) | 2 (3)
Pharyngitis (Infections and infestations) | 0 (0) | 2 (2)
Respiratory Tract Infection (Infections and infestations) | 1 (2) | 0 (0)
Nasopharyngitis (Infections and infestations) | 1 (1) | 1 (1)
Conjunctivitis (Infections and infestations) | 0 (0) | 1 (1)
Gastroenteritis Norovirus (Infections and infestations) | 0 (0) | 1 (1)
Pharyngotonsilitis (Infections and infestations) | 0 (0) | 1 (1)
Scarlet Fever (Infections and infestations) | 0 (0) | 1 (1)
Sinusitis (Infections and infestations) | 0 (0) | 1 (1)
Platelet Count Increased (Investigations) | 0 (0) | 2 (2)
Tonsillar Hypertrophy (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Dehydration (Metabolism and nutrition disorders) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The PI and/or the institution does not have the right to publish or perform presentations, which contain partial or complete summaries, data, results or any other information obtained as a result of this investigation, without prior written authorization by FIDEC.